CLINICAL TRIAL: NCT00504088
Title: Plaque Removal Versus Open Bypass Surgery For Critical Limb Ischemia
Acronym: PROOF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Company decision to halt study
Sponsor: FoxHollow Technologies (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FHT-P-06-003
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2008-08-20 (Estimated); Status verified 2007-08

CONDITIONS: Peripheral Vascular Diseases
Keywords: CLI; Critical Limb Ischemia; PAD; Peripheral Arterial Disease; Artherosclerosis; Leg Pain; Cardiovascular; Artherectomy; Bypass; Peripheral Bypass; PROOF
MeSH Terms: conditions — Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

INTERVENTIONS:
Procedure: Bypass
Procedure: Silverhawk Plaque Excision

SUMMARY:
To compare the outcome of bypass surgery and plaque excision for treatment of critical limb ischemia in the lower limbs

ELIGIBILITY:
Inclusion Criteria:

* Ischemic rest pain for more than 2 weeks or ulceration or gangrene of the foot or toes (Rutherford Becker Category 4, 5 or 6)
* Willing and able, as evaluated by the PI, to provide Informed Consent
* Willing to undergo up to 5 years of clinical follow up visits as scheduled
* Angiographic pattern of infrainguinal disease that can be reasonably managed either by surgery or plaque excision in the first instance
* Reconstitution of at least one patent target tibial segment below the knee which provides run-off to the foot
* The patient must be >18 years of age
* Target lesion(s) is located at or below the level of the superficial femoral artery
* Target lesion(s) is >50% stenosed by quantitative vascular angiography
* Ability to take at least one of the following types of medications: anti- platelet or anti-thrombotic therapy

Exclusion Criteria:

* Patient has cardiac or cardiovascular comorbidities that would make surgery inappropriate
* Patient has terminal or Stage 4 cancer
* Patient has extensive gangrene that requires both a Below-the-Knee amputation and a revascularization procedure
* Previous stent in the target lesion
* Active infection at planned incision site
* The patient is a pregnant woman
* The patient has significant suprainguinal or Common Femoral disease that can not be treated either prior to or during the index procedure
* Target Lesion is a Chronic Total Occlusion (CTO) that is greater than 15cm in length and has severe, continuous calcification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-10

PRIMARY OUTCOMES:
Major amputation-free survival

CONTACTS AND LOCATIONS:
Overall Officials: James F. McKinsey, M.D., Principal Investigator — Columbia University
Locations (31):
- United States (31):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Los Angeles Cardiology/Good Samaritan, Los Angeles, California
  - UC Davis Vascular Center, Sacramento, California
  - San Francisco VA Medical Center, San Francisco, California
  - Stanford University Medical Center/Palo Alto VA, Stanford, California
  - Heart & Vascular Clinic of Northern Colorado, Fort Collins, Colorado
  - Holmes Regional Medical Center, Melbourne, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - University of Chicago, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - St. Vincent, Indianapolis, Indiana
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Vascular Surgery Associates, Baton Rouge, Louisiana
  - Beth Isreal (BIDMC), Boston, Massachusetts
  - St. Vincent Hospital, Worchester, Massachusetts
  - William Beaumont/Southeast Surgical, Royal Oak, Michigan
  - Providence Hospital, Southfield, Michigan
  - University of Mississippi, Jackson, Mississippi
  - Alegent Health Research Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New Mexico Heart Institute, PA, Albuquerque, New Mexico
  - St. Vincent's Medical Center, New York, New York
  - NY Weill Cornell Medical Center, New York, New York
  - Columbia Presbyterian, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland VAMC, Cleveland, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Sentara Heart Hospital, Norfolk, Virginia
  - Madigan Army Medical Center, Tacoma, Washington